CLINICAL TRIAL: NCT05302336
Title: A Randomized Controlled Study of AC (Doxorubicin Hydrochloride Liposome/Cyclophosphamide) vs TC (Docetaxel/Cyclophosphamide) Regimens for Postoperative Adjuvant Chemotherapy in Patients With HR-positive, HER2-negative Early Breast Cancer
Brief Title: AC vs TC in Patients With HR-positive, HER2-negative Early Breast Cancer
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2021-1122
Record Dates: First submitted 2022-03-20; First posted 2022-03-31 (Actual); Last update posted 2022-04-14 (Actual); Status verified 2022-03

CONDITIONS: Breast Cancer; Chemotherapeutic Toxicity
MeSH Terms: conditions — Breast Neoplasms | interventions — liposomal doxorubicin; Cyclophosphamide

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Liposomal doxorubicin + Cyclophosphamide (Active Comparator): Liposomal doxorubicin + cyclophosphamide A 35mg(per r square meter of body surface)+C 600mg(per r square meter of body surface) every 3 weeks for 4 cycles
  Interventions: Drug: Liposomal doxorubicin + Cyclophosphamide vs Docetaxel + Cyclophosphamide
- Docetaxel + Cyclophosphamide (Active Comparator): Docetaxel + Cyclophosphamide T 75mg(per r square meter of body surface)+C 600mg(per r square meter of body surface) every 3 weeks for 4 cycles
  Interventions: Drug: Liposomal doxorubicin + Cyclophosphamide vs Docetaxel + Cyclophosphamide

INTERVENTIONS:
Drug: Liposomal doxorubicin + Cyclophosphamide vs Docetaxel + Cyclophosphamide — All patients who meet the inclusion criteria must first sign the "Informed Consent" after learning about the details of the trial, and they can be formally enrolled only when they have completed all the pre-enrollment examinations and are qualified. Recruitment will continue until the planned number of cases is completed. The trial was not terminated until each surviving patient was followed for at least 60 months after treatment ended or when all patients had died. The randomization table was generated by the SAS software program, and the patients were randomly divided into the experimental group (AC liposomal doxorubicin + cyclophosphamide) and the control group (docetaxel + cyclophosphamide).

SUMMARY:
Anthracycline-paclitaxel sequential combination therapy is the standard regimen for perioperative chemotherapy in breast cancer. The strategy of perioperative chemotherapy is based on breast cancer subtype, i.e. choice of chemotherapy regimen and hormone receptor (HR) [estrogen receptor and/or progesterone receptor], human epidermal growth factor receptor 2 (HER2) related. Although HR-positive breast cancer has a better prognosis than other subtypes, standard chemotherapy for HR-positive breast cancer has not been established. The American Oncology Research Trial 9735 demonstrated that docetaxel + cyclophosphamide (TC) produced better results than doxorubicin + cyclophosphamide (AC) in adjuvant breast cancer treatment. However, the enrolled subjects of the 9735 trial did not strictly limit the tumor size, and the tumor size of some patients was greater than 5 cm; the hormone status of the patients was not limited, about 1/3 of the patients were ER negative, and the HER-2 status of the patients was not limited; 9735 Half of the trial's enrolled population had axillary lymph node metastases. From a large number of clinical studies, it has been found that the patient's tumor size, ER negative, HER-2 positive, lymph node metastasis and other factors are risk factors for breast cancer recurrence and metastasis after surgery. Therefore, for HR-positive, HER-2-negative early breast cancer patients, whether the TC regimen is superior to the AC regimen remains uncertain. The current CSCO breast cancer treatment still recommends the AC regimen as one of the options for adjuvant breast cancer treatment. Other studies have shown a benefit of anthracyclines in high-risk HR-positive disease, and TC is a suitable option for lower risk. The TC regimen had a higher incidence of myelosuppression and allergy than the AC regimen.

DETAILED DESCRIPTION:
At present, the liposomal doxorubicin developed on the basis of doxorubicin has been used for the first-line treatment of advanced breast cancer, and both NCCN and CSCO guidelines have related recommendations. However, the application of liposomal doxorubicin in adjuvant therapy of breast cancer still lacks sufficient evidence-based medicine. The current research shows that doxorubicin under the encapsulation of liposomes prolongs the half-life of the drug, reduces the cardiotoxicity, and the drug is continuously enriched in the tumor tissue to improve the anti-tumor activity. In addition, liposomal doxorubicin has the advantage of less hair loss during chemotherapy, which meets the needs of some clinical patients for hair protection. There is still a lack of clinical studies on the use of AC (liposomal doxorubicin/cyclophosphamide) with other early breast cancer adjuvant chemotherapy regimens. This study aimed to evaluate the efficacy and safety of AC (liposomal doxorubicin + cyclophosphamide) and TC (docetaxel + cyclophosphamide) regimens as adjuvant therapy for HR+ HER2- early breast cancer.

ELIGIBILITY:
Inclusion Criteria:

1. Age: 18~70 years old, female;
2. Patients with primary breast cancer diagnosed by histopathology and clinical stage of T1b-2 N0;
3. The expression of HER-2 is negative by immunohistochemistry (IHC). If the expression of HER-2 is 2+, in situ hybridization is required to confirm that the HER-2 gene is not amplified; HR+.
4. ECOG physical fitness score 0-1 points;
5. LVEF≥55%;
6. Bone marrow function: neutrophils≥1.5×109/L, platelets≥100×109/L, hemoglobin≥90g/L;
7. Liver and kidney function: serum creatinine ≤1.5 times the upper limit of normal; AST and ALT ≤2.5 times the upper limit of normal; total bilirubin ≤1.5 times the upper limit of normal, or ≤2.5 times the upper limit of normal when the patient has Gilbert's syndrome ;
8. The patient has good compliance with the planned treatment, can understand the research process of this study and sign the written informed consent.

Exclusion Criteria:

1. Received cytotoxic chemotherapy, endocrine therapy, biological therapy or radiation therapy for any reason;
2. New York Heart Association (NYHA) score identifies patients with heart disease of grade II or above (including grade II);
3. Patients with severe systemic infection or other serious diseases;
4. Patients who are known to be allergic or intolerant to chemotherapy drugs or their excipients;
5. Other malignant tumors have occurred in the past 5 years, except for skin cancer of cured cervical carcinoma in situ and non-melanoma;
6. Patients of childbearing age who are pregnant or breastfeeding and who refuse to take appropriate contraceptive measures during this trial;
7. Participated in other experimental studies within 30 days before the administration of the first dose of the investigational drug;
8. Patients judged by the investigator to be inappropriate to participate in this study.

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 402 (Estimated)
Dates: Start 2022-05-01 (Estimated); Primary Completion 2024-12-30 (Estimated); Study Completion 2024-12-30 (Estimated)

PRIMARY OUTCOMES:
disease-free survival | 5 years
  the length of time after primary treatment for a cancer ends that the patient survives without any signs or symptoms of that cancer

SECONDARY OUTCOMES:
side effect | 1 year
  hair loss: Sinclair scale for the female pattern was used to evaluate hair loss. Stage 1 is normal. Stage 2 shows the widening of the central part. Stage 3 shows a widening of the central part and loss of volume lateral to the part line. Stage 4 shows the development of a bald spot anteriorly. Stage 5 shows advanced hair loss. Hair loss was assessed after the second and fourth chemotherapy treatments.

CONTACTS AND LOCATIONS:
Locations (1):
- Second Affiliated Hospital, School of Medicine, Zhejiang University, China, Hanzhou, Zhejing, China

IPD SHARING:
Plan to Share IPD: No